CLINICAL TRIAL: NCT02608541
Title: Sheffield Multiple Rib Fractures Study: Evolution of Classification, Management and Outcomes
Brief Title: Sheffield Multiple Rib Fractures Study:
Acronym: SMuRFS
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH19022; 183712 (Other: IRAS)
Record Dates: First submitted 2015-10-12; First posted 2015-11-18 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2017-12

CONDITIONS: Rib Fractures
Keywords: Multiple Rib Fractures, Frail Chest
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective rib fracture fixation: patients presenting since 2006 with multiple rib fractures or flail chest, managed operatively or non-operatively
  Interventions: Other: rib fracture fixation
- Prospective rib fracture fixation: patients presenting from October 2015 to October 2017 with multiple rib fractures or flail chest, managed operatively or non-operatively
  Interventions: Other: rib fracture fixation

INTERVENTIONS:
Other: rib fracture fixation — Use of MatrixRib, where indicated, according to departmental protocol

SUMMARY:
An observational study to derive clinically relevant and predictive rib fracture classification systems, based on retrospective and prospective cohorts, incorporating assessment of PROMs (Patient Reported Outcome Measures) and healthcare utilisation

DETAILED DESCRIPTION:
The aim of this study is to derive radiology-based classifications of rib fractures and to test whether such classifications have a value in the prediction of clinical outcomes and patient reported outcome measures. The first aspect of work is to analyse existing radiology investigations (plain chest radiography (CXR) and derive classifications of rib fractures that, in the retrospective cohort of operated and non-operated cases, could have potential value in the guidance of management and prediction of clinical outcomes. The second aspect will be to evaluate the feasibility of collection of Patient Reported Outcome Measures in patients suffering multiple rib fractures, which will be used to assess the impact of the radiological classifications. The indications for surgery will remain according to current clinical practice and the management algorithms that have been developed previously in the department.

ELIGIBILITY:
Inclusion Criteria:

* Multiple simple rib fractures
* Flail chest

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple rib fractures (+/- flail chest) presenting to Sheffield Major Trauma Centre or the surrounding Trauma Units
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Acute Pain | up to 2 years
  Visual Analogue Score

SECONDARY OUTCOMES:
Forced Expired Volume in 1 second (FEV1) | up to 2 years
Forced Vital Capacity (FVC) | up to 2 years
Length of critical care unit stay | up to 1 year
Complications during critical care unit stay | up to 1 year
  adverse events as assessed by CTCAE v4.0
Length of hospital stay | up to 1 year
Complications during hospital stay | up to 1 year
  adverse events as assessed by CTCAE v4.0
Quality of Life - SF36 (Short Form 36) | up to 2 years
  SF-36
Quality of Life - EQ5D | up to 2 years
  EuroQol Group EQ5D
Quality of Life - EORTC (European Organisation for the Research and Treatment of Cancer) QLQ-C30 (Quality of Life Questionnaire - Cancer-30) | up to 2 years
  EORTC QLQ-C30
Quality of Life - EORTC QLQ-LC13 (Lung Cancer13) | up to 2 years
  EORTC QLQ-LC13
Healthcare cost | up to 2 years
  procedural costs plus hospital cost plus community healthcare costs

CONTACTS AND LOCATIONS:
Overall Officials: John G Edwards, FRCS(C/Th), Study Chair — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom